CLINICAL TRIAL: NCT03709277
Title: Patient-tailored Interventions to Improve Specialty Medication Adherence: Results From a Prospective Randomized Controlled Trial
Brief Title: Interventions to Improve Specialty Medication Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Amanda Kibbons, Clinical Pharmacist, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 181452
Record Dates: First submitted 2018-10-11; First posted 2018-10-17 (Actual); Results first posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Adherence, Medication; Nonadherence, Medication
Keywords: Specialty; Pharmacist Intervention
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacist-Driven Intervention (Experimental): The study group will receive a patient-tailored, pharmacist-driven intervention(s) to overcome patient-specific barriers to adherence. Each patient in the study group will be intervened upon using a protocol that is based on their reason for non-adherence.
  Interventions: Behavioral: Pharmacist-Driven Intervention
- Standard of Care (No Intervention): The usual care group will receive the standard of care provided to all patients that utilize Vanderbilt Specialty Pharmacy.

INTERVENTIONS:
Behavioral: Pharmacist-Driven Intervention — The pharmacist will investigate patient assistance options for patients who cannot afford their specialty medication, reach out to prescribers when needed to address intolerance/adverse effects, improve health literacy, recommend options for forgetfulness, make every effort to reach patient, address clinical and financial barriers to unresponsiveness (lack of lab completion, not returning to clinic, etc.)
  Arms: Pharmacist-Driven Intervention

SUMMARY:
Patients deemed nonadherent to their specialty medications will be randomized to receive 8 months of patient-tailored adherence interventions and follow up from a specialty pharmacist as needed or the standard of care. Medication adherence will be measured using proportion of days covered (PDC) at 8-months post-randomization to determine if the intervention improved specialty medication adherence.

DETAILED DESCRIPTION:
This will be a single-center, prospective, randomized controlled trial. A report of patients who use the Vanderbilt Specialty Pharmacy (VSP) will be generated daily for patients with a proportion of days covered (PDC) < 90% in the previous 4 and 12 months based on pharmacy claims. Patients who meet criteria will be randomized to receive an intervention corresponding to their specific reason for nonadherence and follow up from a specialty pharmacist or to receive usual care. For patients who are randomized to receive an intervention, the specialty pharmacist will review their medication fill history and electronic health record to identify potential reasons for nonadherence or to see if the pharmacy claims inappropriately categorized them as nonadherent (this could be due to holding treatment for a clinical reason, transferring the prescription outside of VSP or other reasons listed in Table 2). After reviewing the patient's pharmacy and medical history, if the pharmacist believes they are truly nonadherent (not taking medication as prescribed), the patient will be contacted to identify potential reasons for nonadherence and intervention(s) will be provided to combat the identified reasons for nonadherence. Adherence rates for those receiving the additional adherence interventions and those receiving standard of care will be calculated 8 months after the date of randomization. The reasons for nonadherence and the intervention to improve adherence rates will be documented in a secured REDCap database. It is important to note that the adherence pharmacist is not study staff, but a full-time employee of the health-system specialty pharmacy performing normal specialty pharmacist functions. The randomization to receive these services or not will allow for evaluation of their efficacy.

ELIGIBILITY:
Inclusion Criteria:

* The same medication (at the Generic Product Identifier level 12) filled ≥4 times in the 12 months before date of import into the study database
* Prescription generated from one of the following Vanderbilt outpatient specialty clinics: Pediatric Rheumatology, Pediatric Gastroenterology/Inflammatory Bowel Disease, adult Vanderbilt Rheumatology clinics, Dermatology, Hematology, Adult Endocrinology, Neurology, Asthma Sinus & Allergy, Idiopathic Pulmonary Fibrosis, Pulmonary Arterial Hypertension, Cystic Fibrosis, Multiple Sclerosis, Neurology, or a Lipid clinic
* Proportion of Days Covered (PDC) < 90% over the previous 4 months and 12 months

Exclusion Criteria:

* Prescription issued by a non-VUMC provider
* Planned treatment discontinuation in the subsequent eight months
* More than one unique specialty medication from the same clinic in the previous four months
* Patients with > 30 gap days in the previous four months and whose last fill was > 30 days from importing into the study database.
* Any reason for misidentified nonadherence in the previous four months
* Deceased patients
* Incarcerated patients

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2022-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Autumn D Zuckerman, Pharm.D., Study Director — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared

REFERENCES:
- [Background] Iuga AO, McGuire MJ. Adherence and health care costs. Risk Manag Healthc Policy. 2014 Feb 20;7:35-44. doi: 10.2147/RMHP.S19801. eCollection 2014. PMID 24591853
- [Background] Brown MT, Bussell JK. Medication adherence: WHO cares? Mayo Clin Proc. 2011 Apr;86(4):304-14. doi: 10.4065/mcp.2010.0575. Epub 2011 Mar 9. PMID 21389250
- [Background] Tan H, Cai Q, Agarwal S, Stephenson JJ, Kamat S. Impact of adherence to disease-modifying therapies on clinical and economic outcomes among patients with multiple sclerosis. Adv Ther. 2011 Jan;28(1):51-61. doi: 10.1007/s12325-010-0093-7. Epub 2010 Dec 6. PMID 21153000
- [Background] Jabbour EJ, Kantarjian H, Eliasson L, Cornelison AM, Marin D. Patient adherence to tyrosine kinase inhibitor therapy in chronic myeloid leukemia. Am J Hematol. 2012 Jul;87(7):687-91. doi: 10.1002/ajh.23180. Epub 2012 Mar 31. PMID 22473898
- [Background] Koncz T, Pentek M, Brodszky V, Ersek K, Orlewska E, Gulacsi L. Adherence to biologic DMARD therapies in rheumatoid arthritis. Expert Opin Biol Ther. 2010 Sep;10(9):1367-78. doi: 10.1517/14712598.2010.510508. PMID 20681888
- [Background] Butt AA, Yan P, Shaikh OS, Chung RT, Sherman KE; ERCHIVES study. Treatment adherence and virological response rates in hepatitis C virus infected persons treated with sofosbuvir-based regimens: results from ERCHIVES. Liver Int. 2016 Sep;36(9):1275-83. doi: 10.1111/liv.13103. Epub 2016 Mar 24. PMID 26928927
- [Background] Andrade SE, Kahler KH, Frech F, Chan KA. Methods for evaluation of medication adherence and persistence using automated databases. Pharmacoepidemiol Drug Saf. 2006 Aug;15(8):565-74; discussion 575-7. doi: 10.1002/pds.1230. PMID 16514590
- [Derived] Kibbons AM, Peter M, DeClercq J, Choi L, Bell J, Jolly J, Cherry E, Alhashemi B, Shah NB, Zuckerman AD. Pharmacist Interventions to Improve Specialty Medication Adherence: Study Protocol for a Randomized Controlled Trial. Drugs Real World Outcomes. 2020 Sep 21:1-11. doi: 10.1007/s40801-020-00213-8. Online ahead of print. PMID 32983839
- [Derived] Kibbons AM, Peter M, DeClercq J, Choi L, Bell J, Jolly J, Cherry E, Alhashemi B, Shah NB, Zuckerman AD. Pharmacist Interventions to Improve Specialty Medication Adherence: Study Protocol for a Randomized Controlled Trial. Drugs Real World Outcomes. 2020 Dec;7(4):295-305. doi: 10.1007/s40801-020-00213-8. PMID 32955714
- See also: Update on Medication Quality Measures in Medicare Part D Plan Star Ratings-2018 — https://q1medicare.com/PartD-2018StarRatingOverallPlanQuality.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Patient-tailored Intervention: The study group will receive a patient-tailored intervention(s) to overcome their specific barrier(s) to adherence. Each patient in the study group will be intervened upon using a protocol that is based on their reason for non-adherence and follow up will continue until 8 months post-enrollment.
  Pharmacist-Driven Intervention: The pharmacist will provide instructions for setting up phone reminders, investigate patient assistance options, reach out to prescribers to address intolerance/adverse effects, provide medication counseling and/or written materials, make every effort to reach patients for refills, address clinical and financial barriers to unresponsiveness (lack of lab completion, not returning to clinic, etc.)
- Standard of Care: The Standard of Care Group will receive the standard of care provided to all patients that utilize Vanderbilt Specialty Pharmacy.
Period: Overall Study
Arm/Group | Patient-tailored Intervention | Standard of Care
Started | 218 | 220
Completed | 218 | 220
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 438 patients were randomized (218 to intervention and 220 to usual care). Reasons for nonadherence in the intervention arm are from all 218 patients. Baseline demographics include all randomized patients; however, the analysis only includes randomized patients with at least 2 fills in the 8 months post-enrollment (199 usual care and 201 intervention)
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient-tailored Intervention | Standard of Care | Total
Number analyzed (Participants) | 218 | 220 | 438
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54 [40 to 63] | 54 [41 to 65] | 54 [40 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155 | 143 | 298
  Male | 63 | 77 | 140
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 34 | 59
  White | 186 | 174 | 360
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 12 | 19
Region of Enrollment [Number; unit: participants]
  United States | 218 | 220 | 438
Median 12-month baseline proportion of days covered (PDC) [Median (Inter-Quartile Range); unit: proportion of days covered (PDC)] | 0.88 [0.78 to 0.90] | 0.86 [0.78 to 0.89] | 0.87 [0.78 to 0.90]

OUTCOME MEASURES:

1. Primary Outcome: Median Proportion of Days Covered (PDC) at 8-months Post-enrollment
Description: Proportion of days covered (PDC) is a calculated value ranging from 0 to 1 where 1 indicates 100% adherence to medication and 0 indicates zero adherence to medication. It uses a patient's refill history to calculate the days' supply obtained over a time period (in days) divided by the time period (in days). It requires at least 2 refills.
Time Frame: 8 months post-enrollment
Population: Only patients with at least 2 fills after their enrollment date were analyzed due to PDC calculations requiring at least 2 fills. Of the 218 patients in the intervention arm, 201 were analyzed. Of the 220 usual care patients, 199 were analyzed.
Measure: Median (Inter-Quartile Range); unit: proportion of days covered (PDC)
Groups:
- Patient-tailored Intervention: The Intervention arm will receive a patient-tailored intervention(s) to overcome their specific barrier(s) to adherence. Each patient in the study group will be intervened upon using a protocol that is based on their reason for non-adherence and follow up will continue until 8 months post-enrollment.
  Pharmacist-Driven Intervention: The pharmacist will provide instructions for setting up phone reminders, investigate patient assistance options, reach out to prescribers to address intolerance/adverse effects, provide medication counseling and/or written materials, make every effort to reach patients for refills, address clinical and financial barriers to unresponsiveness (lack of lab completion, not returning to clinic, etc.)
- Usual Care: The Usual care arm will receive the standard of care provided to all patients that utilize Vanderbilt Specialty Pharmacy.
Arm/Group | Patient-tailored Intervention | Usual Care
Number analyzed (Participants) | 201 | 199
proportion of days covered (PDC) | 0.94 [0.84 to 1.0] | 0.88 [0.75 to 0.97]
Statistical Analysis 1: Comparison: Patient-tailored Intervention vs Usual Care; Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Median Proportion of Days Covered (PDC) at 6-months Post-enrollment
Description: as for outcome 1
Time Frame: 6 months post-enrollment
Population: Only patients with at least 2 fills after their enrollment date were analyzed due to PDC calculations requiring at least 2 fills. Of the 218 patients in the intervention arm, 201 were analyzed. Of the 220 usual care patients, 195 were analyzed.
Measure: Median (Inter-Quartile Range); unit: Proportion of days covered (PDC)
Arm/Group | Patient-tailored Intervention | Usual Care
Number analyzed (Participants) | 201 | 195
Proportion of days covered (PDC) | 0.95 [0.84 to 1.00] | 0.90 [0.76 to 0.98]
Statistical Analysis 1: Comparison: Patient-tailored Intervention vs Usual Care; Test type: Superiority; p = 0.003, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Reasons for Nonadherence in the Intervention Arm
Description: Reasons for nonadherence were obtained from a combination of electronic health records and patient-reported reasons. Since only intervention patients were contacted during this study, only reasons from the intervention arm are reported. Reasons were collected for each patient starting on the date of enrollment until 8-months post-enrollment starting from the date the study began (May 2019) until the study was complete (April 2022).
Time Frame: 35 months
Population: Reasons for nonadherence were provided for all 218 patients randomized to the intervention arm (not just for the patients included in the analysis). Patients may have had more than one reason. Reasons for nonadherence were not collected for the usual care arm as the specialty pharmacist had no contact with the usual care patients.
Measure: Number; unit: Reasons
Groups:
- Intervention Arm: Reasons for nonadherence in the intervention arm
Arm/Group | Intervention Arm
Number analyzed (Participants) | 218
Reasons
  Memory | 81
  Unreachable for refill | 60
  No known reason | 35
  Unresponsive to refill requirements | 31
  Clinical | 25
  Social issues | 23
  Health literacy | 19
  Health system error | 15
  Financial | 8

4. Secondary Outcome: Median Proportion of Days Covered (PDC) at 12-months Post-enrollment
Description: as for outcome 1
Time Frame: 12 months post-enrollment
Population: Only patients with at least 2 fills after their enrollment date were analyzed due to PDC calculations requiring at least 2 fills. Of the 218 patients in the intervention arm, 201 were analyzed. Of the 220 usual care patients, 200 were analyzed.
Measure: Median (Inter-Quartile Range); unit: Proportion of days covered (PDC)
Arm/Group | Patient-tailored Intervention | Usual Care
Number analyzed (Participants) | 201 | 200
Proportion of days covered (PDC) | 0.93 [0.82 to 0.98] | 0.87 [0.72 to 0.95]
Statistical Analysis 1: Comparison: Patient-tailored Intervention vs Usual Care; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were not assessed
Description: All-Cause Mortality, Serious, and other (not including serious) Adverse Events were not monitored/assessed.
Arm/Group | Patient-tailored Intervention | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-09-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT03709277/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-17): https://cdn.clinicaltrials.gov/large-docs/77/NCT03709277/SAP_001.pdf